CLINICAL TRIAL: NCT07320833
Title: Postoperative Analgesic Efficacy of Ultrasound Guided Para-sartorial Compartments (PASC) Block Versus Combined Femoral-Sciatic Nerve Block in Patients Undergoing Total Knee Arthroplasty: A Double-Blind Randomized Comparative Study
Brief Title: Ultrasound-Guided PASC Block vs Femoral-Sciatic Nerve Block for Postoperative Analgesia After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Elsayed Seif, Resident of Anesthesia, Intensive Care and Pain Management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MD 29/2023
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis; Postoperative Pain; Total Knee Arthroplasty
Keywords: Total knee arthroplasty (TKA); Total knee replacement (TKR); Para-sartorial compartments (PASC) block; Femoral nerve block; Sciatic nerve block; Ultrasound-guided nerve block; Regional anesthesia; Multimodal analgesia; Nalbuphine rescue analgesia; Numeric Rating Scale (NRS); Modified Bromage scale
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, two-arm parallel-group trial comparing ultrasound-guided PASC block versus combined ultrasound-guided femoral-sciatic nerve block for postoperative analgesia and motor function after total knee arthroplasty.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are unaware of group assignment. Outcome data are collected by an anesthesiologist blinded to the performed block technique. The anesthesiologist performing the block is not involved in postoperative assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Nerve Block plus Sciatic Nerve Block (Active Comparator): After induction of general anesthesia, participants receive an ultrasound-guided single-shot femoral nerve block with 15 milliliters of 0.25% bupivacaine and an ultrasound-guided single-shot popliteal sciatic nerve block with 15 milliliters of 0.25% bupivacaine. Postoperative multimodal analgesia includes intravenous acetaminophen and ketorolac. Rescue analgesia is intravenous nalbuphine 5 milligrams when the Numeric Rating Scale pain score is 3 or higher, up to 20 milligrams per day.
  Interventions: Procedure: Ultrasound-Guided Femoral Nerve Block plus Sciatic Nerve Block
- Para-sartorial Compartments Block (Experimental): After induction of general anesthesia, participants receive an ultrasound-guided single-shot para-sartorial compartments block using a single needle entry point with three injections of 0.25% bupivacaine: 10 milliliters inside the femoral triangle with periarterial and subsartorial spread, 10 milliliters in the subsartorial plane at the apex of the femoral triangle between sartorius and vastus medialis muscles, and 10 milliliters in the suprasartorial compartment at the level of the intermediate femoral cutaneous nerve (total 30 milliliters). Postoperative multimodal analgesia includes intravenous acetaminophen and ketorolac. Rescue analgesia is intravenous nalbuphine 5 milligrams when the Numeric Rating Scale pain score is 3 or higher, up to 20 milligrams per day.
  Interventions: Procedure: Ultrasound-Guided Para-sartorial Compartments Block

INTERVENTIONS:
Procedure: Ultrasound-Guided Femoral Nerve Block plus Sciatic Nerve Block — Single-shot ultrasound-guided femoral nerve block (15 milliliters of 0.25% bupivacaine) plus single-shot ultrasound-guided popliteal sciatic nerve block (15 milliliters of 0.25% bupivacaine), performed after induction of general anesthesia using sterile technique.
  Arms: Femoral Nerve Block plus Sciatic Nerve Block
Procedure: Ultrasound-Guided Para-sartorial Compartments Block — Single-shot ultrasound-guided para-sartorial compartments block performed after induction of general anesthesia using a single needle entry point and three injections of 0.25% bupivacaine: 10 milliliters in the femoral triangle with periarterial and subsartorial spread, 10 milliliters in the subsartorial plane at the apex of the femoral triangle, and 10 milliliters in the suprasartorial compartment at the level of the intermediate femoral cutaneous nerve (total 30 milliliters).
  Arms: Para-sartorial Compartments Block

SUMMARY:
This randomized, double-blind comparative study evaluates postoperative analgesic efficacy and motor effects of ultrasound-guided para-sartorial compartments (PASC) block versus ultrasound-guided combined femoral-sciatic nerve block in patients undergoing total knee arthroplasty. The primary endpoint is total nalbuphine rescue analgesia consumption in the first 24 postoperative hours. Secondary endpoints include pain scores (NRS), motor function using a modified Bromage scale, block performance characteristics, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 to 70 years
* Scheduled for elective total knee arthroplasty under general anesthesia
* American Society of Anesthesiologists physical status class I or II
* Provided written informed consent

Exclusion Criteria:

* American Society of Anesthesiologists physical status class III or IV
* Pre-existing neurological abnormality of the lower extremity
* Infection near the planned block site
* History of psychiatric illness
* History of drug abuse
* Known allergy to local anesthetics or any study medications (bupivacaine, acetaminophen, ketorolac, nalbuphine)

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Total Rescue Analgesia Requirement (Nalbuphine) | First 24 hours after surgery.
  Total dose of intravenous nalbuphine (in milligrams) administered as rescue analgesia when the Numeric Rating Scale pain score is 3 or higher, with a maximum daily dose of 20 milligrams.

SECONDARY OUTCOMES:
Postoperative Pain Intensity (Numeric Rating Scale) | 30 minutes after admission to the post-anesthesia care unit, and 3 hours, 6 hours, 12 hours, and 24 hours after surgery.
  Pain intensity measured using the Numeric Rating Scale (0 = no pain, 10 = worst possible pain).
Motor Block Assessment (Modified Bromage Scale) | 2 hours, 4 hours, 6 hours, 12 hours, 18 hours, and 24 hours after surgery.
  Motor function assessed using the modified Bromage scale: 1 = complete block (unable to move knee or feet), 2 = almost complete (able to move feet only), 3 = partial (just able to move knees), 4 = none (full flexion of knees and feet).
Block Performance Time | During block performance immediately after induction of general anesthesia.
  Time from ultrasound scanning start to completion of local anesthetic injection (in minutes).
Block Duration | Up to 24 hours after surgery.
  Duration of sensory and motor effects of the nerve block as assessed clinically (in hours).
Postoperative Nausea | First 24 hours after surgery.
  Presence of postoperative nausea during the first postoperative day.
Postoperative Vomiting | First 24 hours after surgery.
  Presence of postoperative vomiting during the first postoperative day.
Sedation (Richmond Agitation-Sedation Scale) | First 24 hours after surgery.
  Richmond Agitation-Sedation Scale score ranging from +4 (combative) to -5 (unarousable); 0 indicates alert and calm.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the primary and secondary outcomes (including total nalbuphine rescue dose, Numeric Rating Scale pain scores, modified Bromage motor scores, procedure time, block duration, and adverse events) will be made available to qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the primary manuscript and will remain available for 5 years.
Access Criteria: Requests should include a brief proposal and analysis plan. Access will be provided after review and approval by the study investigators and completion of a data use agreement. Data will be shared in a de-identified format.